CLINICAL TRIAL: NCT06979349
Title: Respiratory Muscle Strength, Respiratory Muscle Endurance, Cough Strength and Balance in Adolescent Volleyball Players
Brief Title: Respiration and Balance in Adolescent Volleyball Players
Status: Recruiting | Type: Observational
Sponsor: Izmir Democracy University (Other)
Responsible Party: Principal Investigator, Gulsah Bargi, Assoc. Prof. Dr., Izmir Democracy University
Other Study IDs: Adolescent Volleyball Players
Record Dates: First submitted 2025-05-16; First posted 2025-05-18 (Actual); Last update posted 2025-05-18 (Actual); Status verified 2025-05

CONDITIONS: Adolescent Behavior; Athletic Injuries
Keywords: adolescent; volleyball; respiratory muscle; cough; balance
MeSH Terms: conditions — Adolescent Behavior; Athletic Injuries; Cough

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Adolescent Volleyball Players: The group consists of volleyball players who have been actively playing volleyball for at least 1 year and between the ages of 10 and 19
  Interventions: Other: Physical Evaluations in Players

INTERVENTIONS:
Other: Physical Evaluations in Players — Respiratory muscle strength, respiratory muscle endurance, cough strength or balance will be evaluated in adolescent volleyball players.

SUMMARY:
A volleyball player with high respiratory muscle endurance can perform at a high level of efficiency during competitions without experiencing fatigue. However, no study has been found in the literature examining respiratory muscle strength, respiratory muscle endurance, cough strength and balance parameters in adolescent volleyball players which was therefore aimed to investigate the potential relationship between these parameters in this study.

DETAILED DESCRIPTION:
Professional sports performance in adolescent volleyball players who have not yet completed their developmental period may be affected in terms of respiratory muscle strength and endurance, cough strength and balance. However, no study has been found in the literature investigating the relationship between respiratory muscle strength, respiratory muscle endurance, cough strength and balance in adolescent volleyball players and these parameters. Therefore, the aim of our study is to determine the relationship between respiratory muscle strength, respiratory muscle endurance, cough strength and balance in adolescent volleyball players.

ELIGIBILITY:
Inclusion Criteria:

* Being between the ages of 10-19
* Being actively involved in volleyball for at least 1 year
* Voluntarily agreeing to participate in the study
* Volleyball player's parent approving participation in the study

Exclusion Criteria:

* Have been admitted to hospital with a musculoskeletal injury in the last 3 months
* Have any known neurological, orthopedic, rheumatic, and/or cardiovascular disease
* Have been involved in a sport other than volleyball for at least 1 year

Ages: 10 Years to 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Adolescent Volleyball Players consist of research group.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2024-08-10 (Actual); Primary Completion 2026-08-30 (Estimated); Study Completion 2026-08-30 (Estimated)

PRIMARY OUTCOMES:
Respiratory muscle strength assessment | through study completion, an average of 1 year
  Respiratory muscle strength will be measured using a portable spirometer. The pressure will be recorded during a few seconds of maximal inspiration (Müller maneuver) or expiration (Valsalva maneuver) through the mouth.The high value obtained indicates good muscle strength.

SECONDARY OUTCOMES:
Respiratory muscle endurance assessment | through study completion, an average of 1 year
  The respiratory muscle endurance test at increasing threshold load will be measured using POWERbreathe Wellness® Classic Light Resistance device. If the volleyball player cannot continue the test for 10 minutes, the last pressure value at which he can continue ventilation for 2 minutes will be recorded as the respiratory muscle endurance value. Being able to sustain the test for a long time indicates good respiratory muscle endurance.
Evaluation of Cough Strength | through study completion, an average of 1 year
  The volleyball player's peak cough expiratory flow value will be evaluated using a peak flow meter. The best of at least three repetitions will be recorded. The highest value indicates good cough strength.
Balance Assessment | through study completion, an average of 1 year
  Balance will be assessed using the Functional Reach Test (FUT). Volleyball players will reach forward from the waist to the wall. The highest reach value will be recorded.The highest value indicates good balance.

CONTACTS AND LOCATIONS:
Overall Officials: GÜLŞAH BARGI, Study Director — Izmir Democracy University; ÖZLEM ÇİNAR ÖZDEMİR, Prof Dr, Principal Investigator — Bolu abant İzzet Baysal University; CEMRE GÖRÜNMEZOĞLU, MSc, Principal Investigator — Izmir Democracy University; ELİF YEŞİLAY BÜYÜKDERE, MSc, Principal Investigator — Goztepe Sport Club
Locations (1):
- Izmir Democracy University, Konak, İ̇zmi̇r, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Tiaprapong K, Sirikul A, Krajangmek C, Duangthongkul N, Pandam N, Piya-Amornphan N. Awareness of COVID-19 influences on the wellness of Thai health professional students: An ambulatory assessment during the early "new normal" informing policy. PLoS One. 2021 Jun 14;16(6):e0252681. doi: 10.1371/journal.pone.0252681. eCollection 2021. PMID 34125868
- [Background] Fink JB. Forced expiratory technique, directed cough, and autogenic drainage. Respir Care. 2007 Sep;52(9):1210-21; discussion 1221-3. PMID 17716387
- [Background] Duncan PW, Weiner DK, Chandler J, Studenski S. Functional reach: a new clinical measure of balance. J Gerontol. 1990 Nov;45(6):M192-7. doi: 10.1093/geronj/45.6.m192. PMID 2229941
- [Background] Celik Z, Guzel NA, Yuksel F, Kafa N. Lung age and respiratory muscle strength in female volleyball players. Rev Assoc Med Bras (1992). 2021 Oct;67(10):1432-1436. doi: 10.1590/1806-9282.20210639. PMID 35018971
- [Background] American Thoracic Society/European Respiratory Society. ATS/ERS Statement on respiratory muscle testing. Am J Respir Crit Care Med. 2002 Aug 15;166(4):518-624. doi: 10.1164/rccm.166.4.518. No abstract available. PMID 12186831
- [Background] Bahat G, Tufan A, Ozkaya H, Tufan F, Akpinar TS, Akin S, Bahat Z, Kaya Z, Kiyan E, Erten N, Karan MA. Relation between hand grip strength, respiratory muscle strength and spirometric measures in male nursing home residents. Aging Male. 2014 Sep;17(3):136-40. doi: 10.3109/13685538.2014.936001. Epub 2014 Jul 4. PMID 24993454